CLINICAL TRIAL: NCT06638645
Title: Reasons for Prolonged Hospital Stay After Thoracoscopic Anatomical Lung Resections
Brief Title: Prolonged Hospital Stay After Thoracoscopic Anatomical Lung Resections
Acronym: PROTRACT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Sint-Lucas Brugge (Other)
Responsible Party: Principal Investigator, DienstThoracaleEnVasculaireHeelkunde, Clinical professor, University Hospital, Ghent
Other Study IDs: THE-2024-0246
Record Dates: First submitted 2024-10-01; First posted 2024-10-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Minimally Invasive Surgical Procedures; VATS; RATS Surgery; Pulmonary Lobectomy; Pulmonary Segmentectomy; Air Leakage; Postoperative Complication; Pain Postoperative
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing a minimally invasive anatomical lung resection: Patients undergoing a minimally invasive anatomical lung resection, receiving perioperative care according to the ERAS protocol for Lung Surgery
  Interventions: Procedure: VATS/RATS anatomical lung resection

INTERVENTIONS:
Procedure: VATS/RATS anatomical lung resection — Perioperative care according to the ERAS protocol for lung surgery
  Other Names: VATS lobectomy; RATS lobectomy; VATS segmentectomy; RATS segmentectomy

SUMMARY:
In this study, the reasons for prolonged hospital stay after thoracoscopic (video- or robot-assisted) anatomical lung resections are investigated. Currently, whenever possible, these anatomical lung resections are performed thoracoscopically, as they offer significant improvements in terms of postoperative pain, number of postoperative complications, rehabilitation, tolerance for adjuvant chemotherapy, and length of hospital stay. The development of an 'Enhanced Recovery After Surgery' (ERAS) protocol for lung surgery has further reduced hospital stay and the need for opioids for analgesia. Despite the optimal implementation of the ERAS protocol, there are still patients who need to stay in the hospital longer than the median. The aim of this research is to investigate the reasons for this.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for elective minimally invasive (uniportal or multiportal video- or robot-assisted) anatomical lung resection (lobectomy or segmentectomy)
* Informed consent obtained pre-operatively
* Age 18 years or older

Exclusion Criteria:

* Patients younger than 18 years old
* Traumatic event as indication for lung resection
* Non-anatomical lung resections
* Thoracotomy
* Patients already hospitalized for other pathologies, pre-existent and not related to the lung surgery
* Urgent/emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for thoracoscopic anatomical lung resection. An estimated 136 patients should be included after power calculation
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay (days) | immediately after surgery until hospital discharge (1 week on average), up to 3 months
  The primary objective is to investigate the length of hospital stay of patients undergoing minimally invasive thoracoscopic anatomical lung resection with peri-operative care according to the Enhanced Recovery After Surgery (ERAS) protocol for lung surgery

SECONDARY OUTCOMES:
Reasons for delayed discharge (more than 2 days postoperatively) identified through daily questionnaires and review of medical records. | immediately after surgery until hospital discharge (1 week on average), up to 3 months
  * Postoperative pain (NRS)
  * Postoperative nausea and vomiting (yes/no)
  * Air leak duration (days)
Number, frequency and severity of postoperative complications during hospital stay. | immediately after surgery until hospital discharge (1 week on average), up to 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No